CLINICAL TRIAL: NCT06206941
Title: Assessing Benefits and Harms of Cannabis Use in Patients Treated With Immunotherapy for Cancer: a Prospective Cohort Study
Brief Title: IMmunotherapy: Prospective Assessment of Cannabis Treatment in Cancer
Acronym: IMPACT-C
Status: Recruiting | Type: Observational
Sponsor: State University of New York at Buffalo (Other)
Collaborators: Thomas Jefferson University (Other); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Rebecca Ashare, Associate Professor, State University of New York at Buffalo
Other Study IDs: STUDY0007957
Record Dates: First submitted 2023-12-21; First posted 2024-01-16 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cannabis User: Cancer patients being treated with immunotherapy and using cannabis
- Cannabis non-user: Cancer patients being treated with immunotherapy and not using cannabis

SUMMARY:
The purpose of this research is to assess how patients with cancer being treated with Immune Checkpoint Inhibitors (ICI) manage symptoms related to cancer and/or its treatment. Patients use a variety of ways to manage symptoms including traditional and alternative treatments including cannabis, acupuncture, etc. This research will have an important impact on our knowledge of cancer symptom management, and ultimately improve patient care and safety.

Participants will complete online surveys and 7 days of ecological momentary assessments at 0, 1, 2, 4, 6, 9 and 12 month to compare the cannabis users and non cannabis users symptoms.

DETAILED DESCRIPTION:
Immunotherapy:Prospective Assessment of Cannabis Treatment in Cancer (IMPACT-C) is an observational study to assess the side effect of cancer patients going through immunotherapy treatments. The investigators will use a variety of methods to recruit, including generating reports of potentially eligible patients from institutional registries, reviewing Electronic Medical Records (EMR), approaching patients during their regular outpatient visits, taking referrals from oncology teams, and placing study advertisements at strategic locations of the oncology clinics and Facebook sites. If a potentially eligible patient is interested in the study, the research assistant (RA) will review the eligibility checklist. The consent form will be written in easy-to-understand English and administered during a regular office visit or virtually via video/phone meeting, based on patients' convenience and preference. Once informed consent/HIPAA are completed and eligibility is confirmed, participants will complete Baseline measures (see Measurement Table). Those patients that are eligible for the subset of blood draws will review and sign the amendment.

A research assistant (RA) or study staff will collect self-reported data using video or phone calls at all time points; This method has several advantages, including participant convenience and the RAs' ability to directly enter data into a secure study database, thereby reducing the potential for missing data. Assessments range from 30-60 min per time point. In person visits can be arranged if technology is limited at the cancer centers or University.

Ecological Momentary Assessment (EMA). Daily EMA data will be collected for 7 consecutive days at each assessment timepoint (total of 49 days) using web link or an application (app) that can be loaded onto the patients' smart phone (significantly reducing patient burden). The week of data collection in measurement months (0, 1, 2, 4, 6, 9 and 12) will be randomized across participants. Capturing data at various times throughout the month will allow the investigators to account for potential confounding factors (e.g., patients receiving income at the beginning of the month). The EMA (mEMA; ilumivu, Inc. Or through REDCap and Mosio), provides flexibility in survey creation, alert scheduling, and monitoring of participant compliance. The mEMA platforms time stamps all responses to monitor fidelity, is available for both Android and iphone Oporating System (iOS) phones, and allows recording of responses even when Wi-Fi and cellular signals are lost or turned off (e.g., airplane mode). All de-identified data (linked only to participant ID) are synchronized with a secure server. EMA training and assessment procedures will follow prior and on-going work of the investigators. During the Baseline call (Month 0), participants will be trained on proper use of the EMA and will demonstrate the ability to complete both self-initiated assessments (morning assessment) and device-initiated assessments (alerts sent to participant at random times of day). Study staff will complete regular check-ins to troubleshoot any difficulties with the EMA. To improve adherence and reduce burden, participants will select a 9-hour period during which EMA prompts occur each day (our pilot work indicated that a 12-hour period was too long as many patients reported going to bed early and sleeping late).

EMA Measures include, Morning Assessment (user initiated, 1/day, duration 3-7 minutes, timeframe: previous 24 hours) of questions regarding; Cannabis use,Daily use (yes or no) source, form composition, and quantity, Reason for Cannabis use, Pain, sleep, anxiety, nausea, enjoyment, other (6-item checkboxes),Adverse effects (Dizziness, difficult concentrating, Impaired memory, Fatigue (4-item checkboxes),Other medications (Opioids, benzodiazepines, sleep aids, etc.)

Device-initiated Assessments 3 random alarms, 3/day. Every 3 hours over a 9-hour duration: 2-5 min., timeframe: current) of questions on Cannabis use,use since last assessment (yes or no); quantity, form, composition, reason for use (see above), anxiety (2 randomly selected items from the Patient Reported Outcomes Measurement Information System (PROMIS), Pain, Enjoyment of Life & General Activity function (PEG) scale, adverse effects (AE).

Participants will be asked to complete the morning assessment for 7 consecutive days, within 1 hour of waking. Table 3 shows the items assessed. Device-initiated random assessments will be delivered 3 times per day for 7 consecutive days at each timepoint. The device-initiated prompts will be delivered over 9 hours, beginning 3 hours after the participant's usual wake time and divided into three 3-hour blocks (1 assessment per block and constrained so that each assessment is at least 1 hour apart).

Inflammatory marker assay. A subset of 60 patients (30 cannabis users and 30 cannabis non-users) will have 8 milliliter (ml) blood samples drawn at baseline (prior to initiation of ICI treatment) and months 2, 6, & 12 to assess changes in inflammatory markers. Samples will be collected, processed, and de-identified; serum will be stored locally. At the time of blood draw, we will assess whether cannabis has been used in the past 72 h. All three recruitment sites collect and store blood samples that can be used for future research as part of their master protocols. Thus, if we have difficulty enrolling patients prior to the start of treatment, we will have access to these banked samples. Upon study completion, samples from Oregon Health and Science University and University at Buffalo will be shipped to Sydney Kimmel Cancer Center and analyzed by Co-Investigator Dr. Harshyne's highly experienced immunology lab. Specifically, Luminex multiplex assays use xMAP bead-based technology to simultaneously detect and quantitate multiple secreted proteins including cytokines, chemokines, and growth factors in a single sample. The Luminex® xMAP® technology uses color-coded beads coupled with target-specific antibodies allowing the detection of up to 100 soluble analytes in a single 20 ul sample.

Electronic Medical Record Data. Each site will collect clinical data from routinely conducted labs within +/- 1 month of the following time points: baseline, 1, 2, 4, 6, 9, and 12 months. Data to be collected will include blood draw lab data that is routinely collected on all oncology patients during surveillance and survivorship: comprehensive metabolic panel (CMP; inclusive of renal and liver function as well as blood glucose and albumin), complete blood count (CBC) with differential and all applicable tumor markers associated with the cancer type for each patient. Additionally, any acute, unplanned hospitalizations or Emergency Room visits will be noted, inclusive of the reason for admission. All radiographic scans done +/- 1 month of the time point will be recorded with specific notation of progression or regression of disease documented in report.

The data sources in this study include repeated assessments using EMA, monthly assessment of Patient Reported Outcomes (PROs), patients' EMR, for cancer progression and blood samples for inflammatory markers.

The investigator's goal was to use widely validated common data elements while minimizing patient burden. Thus, the investigators chose psychometrically equivalent brief measures when they were available. Investigators also decreased the administration frequency of measures that did not make sense as serial measures. Investigators quantified completion time based on literature or our previous experience with the measure.

Aim 1. Assess benefits and harms of cannabis use over 12-months. Primary outcomes will be from EMA data; monthly surveys are secondary.

Aim 1a (Benefits): Pain. The 3-item PEG scale (Pain, Enjoyment of life, General activity) was chosen for its brevity and validity. PEG scale has been recommended by the Centers for Disease Control and Prevention (CDC) to assess pain and function and recommended by the Methods, Measurement, and Pain Assessment in Clinical Trials (IMMPACT) group that sets the standards of measurement in pain research. A 30% improvement or difference is considered clinically meaningful. Anxiety. The PROMIS Anxiety (SF4a) will be used to assess anxiety via EMA. These 4 items are also included in the 8-item version used in monthly surveys. Sleep. The PROMIS Sleep Disturbance (SF4a) will be used to assess perceptions of sleep quality, perceived difficulties and concerns with falling or staying asleep, and perceptions of satisfaction with sleep. Additional PROs, considered exploratory, are collected during monthly surveys.

Aim 1b (Harms): The presence of the following 4 adverse effects will be assessed via EMA: dizziness, difficulty concentrating, impaired memory, and fatigue. These items were chosen because these are the most common adverse effects of cannabis, common in cancer and its treatments and our pilot data. The Adverse Reactions to Cannabis Scale (ARCS) assesses for the presence of each reaction while using cannabis (yes/no) and for each endorsed reaction, how distressing it was using a 5-point Likert scale (0=Not at all to 4=Severely distressing). Adverse Effects of ICIs including the identification, grading, and recommendations for managing immune-related and other ICI treatment-related AEs will be extracted from the EMR.8-item Cannabis Use Disorders Identification Test-R (CUDIT-R)(past 6 months) assesses consumption, cannabis related problems, dependence, and psychological consequences. CUDIT-R is secondary because it only applies to patients who use cannabis. Additional outcomes, considered exploratory, are collected during monthly surveys.

Aim 2. Test whether cannabis use over time moderates the associations between a measure of neighborhood disadvantage (Area Deprivation Index) and benefits and harms in Aim 1. The investigators use the Area Deprivation Index (ADI) as a composite indicator of Social Disparity of Health (SDoH). Created by the Health Resources & Services Administration, and adapted and validated to the Census Block Group neighborhood level, the ADI is a widely used measure ranking neighborhoods based on socioeconomic disadvantage. Its composite score combines key indicators of socioeconomic status, such as income, education, employment, and housing quality, and is weighted and standardized to create an overall score for each neighborhood (0-100 percentile), with higher scores indicating a higher degree of disadvantage. Across studies, including studies with persons with cancer, ADI has informed health delivery, access, and policy outcomes, especially for the most disadvantaged neighborhoods. Rationale for ADI: While the investigators considered focusing mainly on race and ethnicity or other measures of socioeconomic disadvantage (e.g., Distressed Community Index), we chose ADI for these reasons: (1) ADI has a greater number of SDoH input variables to inform outcomes;(2) Although we will account for self-reported race and ethnicity in our analyses to identify race-based disparities, investigators propose ADI as it is based on a broader set of SDoH variables that are relevant to our study including neighborhood characteristics that have been associated with access to cannabis dispensaries and other types of health and social access; (3) ADI employs area-level indicators of Social Economic Status (SES) at a small geographic scale (9-digit census tracts vs 5-digit zip code in DCI); and (4) investigators opted not to use individual SES as neighborhood disadvantage has been independently associated with poor health outcomes, regardless of an individual's SES. Data suggest that individuals from low-income backgrounds residing in relatively affluent neighborhoods may exhibit better health outcomes than those living in disadvantaged neighborhoods.

Aim 3 (Exploratory). For a subset of patients (n=60) scheduled to receive ICI therapy as a first-line cancer treatment for non-skin solid malignancies, investigators will longitudinally explore whether cannabis use is associated with markers of (a) disease response or progression; (b) clinical outcomes (Table 5); and (c) key immunological markers from baseline (prior to initiation of ICI treatment) and over 12-months. Most data for Aim 3 will be extracted from the EMR (Table 5). Inflammation assays will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* adult age of 21 years or older
* cancer diagnosis and planning or using immunotherapy treatment,
* pain and spend less than 50% in bed or chair
* fluent in english language

Exclusion Criteria:

* use synthetic cannabis or only use Cannabidiol (CBD)
* non users but used in the past 3 months
* prior immunotherapy, Patients receiving immunosuppressants or organ transplant recipients.
* Patients within 6 months of Hospice care.
* Pain that limits movement to more than 50% of their day in bed or chair

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult cancer patients that are treated or plan to be treated with immunotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient Reported Outcomes Measurement Information System: Pain interference | 0,1,2,4,6,9 and 12 months
  Pain interference with daily life and enjoyment on a 5 item scale of not at all to very much. Higher score indicates worse outcome.
Patient Reported Outcomes Measurement Information System: Sleep | 0,1,2,4,6,9 and 12 months
  PROMISE sleep disturbance on a 5 item scale of not at all to very much. Higher score indicates worse outcome.
Patient Reported Outcomes Measurement Information System:Anxiety | 0,1,2,4,6,9 and 12 months
  Anxiety on a 5 item scale of never to always. Higher score indicates worse outcome. Higher score indicates worse outcome.
Adverse reaction of Cannabis | 0,1,2,4,6,9 and 12 months
  Adverse reaction to Cannabis Scale of present side effects and 5 item scale of how distressing the symptoms were experienced. Higher score indicates worse outcome.
Cannabis Use Disorder Identification Test | 0,1,2,4,6,9 and 12 months
  Cannabis Use Disorder Identification Test (CUDIT), the usage of cannabis and 5 item scale of never to daily or almost daily. Higher score indicates worse outcome.
Patient Reported Outcomes Measurement Information System: Depression | 0,1,2,4,6,9 and 12 months
  Emotional Distress-Depression on a 5 item scale of never to always, level of sexual activity, emotional well-being, functional well-being and additional concerns on a 5 item scale not at all to very much. Higher score indicates worse outcome.
Patient Reported Outcomes Measurement Information System: Cognitive Function | 0,1,2,4,6,9 and 12 months
  Cognitive Function-Abilities on a 5 item scal not at all to very much. Higher score indicates better outcome.
Patient Reported Outcomes Measurement Information System: Fatigue | 0,1,2,4,6,9 and 12 months
  Level of fatigue on a 5 item scale of never to always. Higher score indicates worse outcome.

SECONDARY OUTCOMES:
Quality of Life with cancer | 0,1,2,4,6,9 and 12 months
  Functional Assessment of Cancer Therapy-General. Physical well-being, Social/Family Well being on a 5 item scale of not at all to very much. Higher score indicates worse outcome.
Area Deprivation Index | 0, 2, 6, and 12
  Test cannabis use association with Area Deprivation Index (ADI) and the benefits and harms. The Area Deprivation Index Its composite score combines key indicators of socioeconomic status, such as income, education, employment, and housing quality, and is weighted and standardized to create an overall score for each neighborhood (0-100 percentile), with higher scores indicating a higher degree of disadvantage.

OTHER OUTCOMES:
Immunological markers | 0, 2, 6 and 12 month
  Blood draws to test inflammatory markers. Luminex multiplex assays use xMAP bead-based technology to simultaneously detect and quantitate multiple secreted proteins including cytokines, chemokines, and growth factors in a single sample. The Luminex® xMAP® technology uses color-coded beads coupled with target-specific antibodies allowing the detection of up to 100 soluble analytes in a single 20 ul sample.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Oregon Health and Science University, Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No